CLINICAL TRIAL: NCT02442453
Title: Effect of Scaling and Root Planing Along With Topical Application of Commercially Available Curcuma Longa Gel on Superoxide Dismutase and Malondialdehyde Levels in Saliva of Chronic Periodontitis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tatyasaheb Kore Dental College (Other)
Responsible Party: Principal Investigator, DR.DHANASHREE RAVINDRA AGARWAL, Dr.DHANASHREE RAVINDRA AGARWAL, Tatyasaheb Kore Dental College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DHANASHREE786
Record Dates: First submitted 2015-04-28; First posted 2015-05-13 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- curcuma longa (Active Comparator): curenext gel containing curcuma longa i.e. turmeric has strong antioxidant and antiinflammatory properties.
  Test group:Topical application twice daily for ten minutes after brushing for four weeks.
  Interventions: Drug: Topical application of curenext gel
- Placebo gel (Placebo Comparator): Placebo gel consists of corbopol 934 polymer and triethonalamine. Control group:Topical application twice daily for ten minutes after brushing for four weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Topical application of curenext gel — Topical application of curcuma longa gel along with scaling and root planing in chronic periodontitis subjects
  Other Names: curcuma longa topical gel; curenext gel
  Arms: curcuma longa
Drug: Placebo — Topical application of placebo gel along with scaling and root planing in chronic periodontitis subjects
  Arms: Placebo gel

SUMMARY:
Periodontitis is initiated by microbial biofilm but its progression is mediated by an abnormal host response to biofilm microorganisms.

In a myriad of possible mechanisms that cause periodontal tissue destruction reactive oxygen species (ROS) play an important role. Imbalance between antioxidant defense system of body and ROS lead to a deleterious situation called oxidative stress.

Superoxide dismutase (SOD) is the key enzyme of body's antioxidant defense system whereas malondialdehyde (MDA) is product of lipid peroxidation due to ROS. Free radicals and ROS have short half lives in vivo of 10-6 to 10-9 seconds. Hence measurement of ROS is done by measuring the concentration of biomarkers of tissue destruction.

For treating periodontal disease, conventional mechanical therapy comprising of scaling and root planing (SRP) along with timely maintenance has been a gold standard and any other therapy considered for treating periodontitis should always be used as an adjunctive and never in lieu of it.

Curcumin, a hydrophobic polyphenol, is a principal active constituent of turmeric. Mechanism of action of curcumin is twofold-its role as a strong antioxidant and as a strong antibacterial. Its analgesic, anti-inflammatory and antiseptic properties offer additional benefits.Periodontitis is a chronic disease of oral cavity accompanied by increased oxidative stress. Therefore the clinical application of a natural antioxidant in the form of curcuma longa can be beneficial in reducing oxidative stress and as an adjuvant in treatment of chronic periodontitis.

DETAILED DESCRIPTION:
Aim was to establish efficacy of curcuma longa gel as a topical antioxidant to alleviate oxidative stress associated with chronic periodontitis.The objectives were-1) To evaluate the presence of oxidative stress by biochemical evaluation of SOD levels and free radical damage in the form of MDA levels in whole saliva of chronic periodontitis patients.

2) To show efficacy of curcuma longa gel as topical antioxidant agent on activity of SOD and lipid peroxidation product MDA.

3) To compare SOD and MDA levels after SRP and SRP plus topical application of curcuma longa gel.

4) To compare the clinical parameters such as Plaque index (PI), Gingival index (GI), Sulcus bleeding index (SBI), Probing depth (PD), Clinical attachment level (CAL) between test group (TG) and control group (CG).

ELIGIBILITY:
Inclusion Criteria:

1. Patients within age group of 30 to 55 years.
2. Systemically healthy individuals.
3. Patients with chronic generalized periodontitis (based on American Academy of Periodontology classification 1999).

Exclusion Criteria:

1. Patients with systemic illnesses (i.e., diabetes mellitus, cancer, human immunodeficiency syndrome, bone metabolic diseases, or disorders that compromise wound healing, radiation, or immunosuppressive therapy, xerostomia).
2. Patients on antioxidants, antibiotics and anti-inflammatory drugs.
3. Those receiving periodontal treatment in last six months prior to inception of study
4. History of smoking, tobacco chewing, alcohol consumption.
5. Pregnant and lactating women.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2014-01; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Superoxide dismutase antioxidant enzyme levels in saliva of chronic periodontitis subjetcs | one month